CLINICAL TRIAL: NCT05626868
Title: Intraoperative Abdominal Pressure Measurement in Patients Undergoing Spine Surgeries in Prone Position as a Marker of Renal Damage
Brief Title: Changes of Intra Abdominal Pressure During Surgeries in Prone Position as a Marker of Renal Damage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: MG/M/37/37/20(1)
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Intraabdominal Hypertension; Prone Postion; Spine Surgery
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients for spine surgery in prone position
  Interventions: Device: Intra abdominal pressure measurement

INTERVENTIONS:
Device: Intra abdominal pressure measurement — Device: Biometrix - Intraabdominal pressure monitoring set Intraabdominal pressure monitoring with the intended set in values of milimeters of mercury (mmHg) in real time.

SUMMARY:
Background: Patients undergoing surgical operations in prone position do not have a measure of intra abdominal pressure as a standard procedure. Many of them could have elevated values of this parameter and could be exposed to possible renal damage due to a stiffening of the abdominal muscles while being positioned prone.

Purpose of study: Intraoperative intrabdominal pressure measurement and evaluation of correlation with possible postsurgical complications.

Methodology: Electronic device able to measure intra abdominal pressure is connected between a Foley catheter and a urinary collecting bag. During the procedure, values of the intra abdominal pressure are displayed on a monitor next to anaesthetic machine in real time. The numbers representing the pressure in mmHG are assessed and recorded.

Discussion: Possible correlation between intra abdominal hypertension and postsurgical complications in patients operated in prone position could be a foundation to further clinical trials and presurgical assessment of intraabdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Patients qualified for surgical stabilization of the spine in prone position

Exclusion Criteria:

* No consent to participate in the study or inability to obtain consent
* The inability to insert a urinary catheter
* No indication for urinary catheter
* Patients undergoing palliative treatment
* Patients with advanced liver and kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients qualified for spinal surgery in prone position, who consent to praticipate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase in intra abdominal pressure during surgery. | Intraoperative
  Change in intra abdominal pressure during surgery in prone position.

SECONDARY OUTCOMES:
Correlation of increased abdominal pressure with renal dysfunction assessed by creatinine. | From start to eight hours after the surgery.
  Assessment of renal function in labolatory tests: creatinine change (mg/dl).
Correlation of increased abdominal pressure with renal dysfunction assessed by urea. | From start of surgery to eight hours after the surgery.
  Assessment of renal function in labolatory tests: urea change (mg/dl).
Correlation of increased abdominal pressure with renal dysfunction assessed by potassium. | From start of surgery to eight hours after the surgery.
  Assessment of renal function in labolatory tests: potassium change (mg/dl).
Correlation of increased abdominal pressure with mioglobin. | From start of surgery to eight hours after the surgery.
  Assessment in labolatory tests: mioglobin change (mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kowalczyk, MD, Principal Investigator — Medical Unieveristy of Warsaw
Locations (1):
- Medical University of Warsaw: 1st Department of Anaesthesiology and Intensive Therapy, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No